CLINICAL TRIAL: NCT02613715
Title: Influence of Ethanol in the Bioavailability of Blackberry Juice Anthocyanins in Normal Weight and Overweight/Obese Adults
Brief Title: Bioavailability of Blackberry Juice Anthocyanins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other); Vinoflavo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VINOFLAVO_01
Record Dates: First submitted 2015-11-16; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Overweight and Obesity; Healthy
Keywords: Flavonoids; Anthocyanins; Blackberry Juice; Bioavailability; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blackberry juice with 12% ethanol (Experimental): 250 ml of blackberry juice freshly prepared with 250 g fresh blackberries, 80 ml alcohol beverage (38%) and 17 g sugar.
  Interventions: Dietary Supplement: Blackberry juice with 12% ethanol
- Blackberry juice (Experimental): 250 ml of blackberry juice freshly prepared with 250 g fresh blackberries, 80 ml water and 17 g sugar.
  Interventions: Dietary Supplement: Blackberry juice

INTERVENTIONS:
Dietary Supplement: Blackberry juice with 12% ethanol
  Arms: Blackberry juice with 12% ethanol
Dietary Supplement: Blackberry juice
  Arms: Blackberry juice

SUMMARY:
The main aim of this study is to evaluate the bioavailability of blackberry juice anthocyanins, with or without ethanol, in normal weight and overweight/obese adults.

DETAILED DESCRIPTION:
Anthocyanins (ANT), a particular class of flavonoids that can be found in red wine and red fruits, have been associated with relevant health benefits. It has become clear that the flavonoid bioactive forms in vivo are not necessarily those which occur in nature, but metabolites arising from them after absorption. Therefore, it is important to identify which ANT metabolites are responsible for their health benefits. Since ANT can prevent/treat some of the metabolic features of obesity it is also crucial to study whether ANT bioavailability is not compromised in obesity.

An anthropometric evaluation will allow the classification of subjects according to their body mass index (BMI). A complete medical examination including the assessment of clinical laboratory parameters will also be performed to characterize the health status of recruited subjects.

Before the beginning of the study, the last fecal sample obtained will be collected. Urine samples and peripheral venous blood (10 ml) will be collected from 10 h-fasting subjects. Afterwards, each volunteer will consume 250 ml of blackberry juice with or without ethanol (visit 1 and 2) and blood samples will be collected 15, 30, 60 and 120 min after juice ingestion. Another urine sample will be collected at 120 min. The first fecal sample obtained at least 6 h after juice ingestion will be collected. Blood pressure (0 and 120 min) and glycaemic response (0, 15, 30, 60 and 120 min) will be measured in each visit.

Ethanol was added to the blackberry juice to mimic the concentration presented in red wine (12%).

A thorough screening analysis for ANT will be performed in plasma and urine samples collected from the volunteers at different time points. Fecal samples will also be collected to evaluate the relationship between the presence of ANT metabolites and the gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18-40 years
* BMI>18 kg/m2
* Willing and able to provide written consent

Exclusion Criteria:

* Subjects with current or previous CVD, diabetes or other severe chronic disease
* Subjects under prescription of any chronic medication
* Pregnant or breast-feeding subjects
* Intake of antibiotics in the last 3 months prior to the beginning of the intervention
* Intake of red fruits or red wine in the last 24 h prior to the beginning of the intervention
* Subjects involved in any clinical or food study within the preceding month
* Subjects with a diagnosis of any digestive disease including functional bowel disorder such as IBS

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of anthocyanins and anthocyanins metabolites | At baseline and 15, 30, 60 and 120 minutes after juices consumption

SECONDARY OUTCOMES:
Urinary concentrations of anthocyanins and anthocyanins metabolites | At baseline and 120 minutes after juices consumption
Fecal concentrations of anthocyanins and anthocyanins metabolites | At baseline and at least 6 h after juices consumption
Number of copies of bacterias presented in fecal samples | At baseline and at least 6 h after juices consumption
Blood pressure measured in the left upper arm using an automatic blood pressure monitor | At baseline and 120 minutes after juices consumption
Capillary blood glucose concentration | At baseline and 15, 30, 60 and 120 minutes after juices consumption

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — CINTESIS - Faculty of Medicine of University of Porto
Locations (1):
- CINTESIS - Faculty of Medicine of the University of Porto, Porto, Portugal